CLINICAL TRIAL: NCT06755827
Title: Emotion Regulation Intervention to Improve Neural Responsiveness and Health
Brief Title: Pilot Testing a Novel Approach to Pediatric Obesity Treatment
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Caroline Cummings, PhD, Assistant Professor, Texas Tech University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-0493; U24DK132740 (NIH)
Record Dates: First submitted 2024-12-17; First posted 2025-01-01 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Overweight Adolescents; Obese Adolescents
Keywords: overweight; obesity; adolescents; neuronal responsiveness; emotion regulation
MeSH Terms: conditions — Overweight; Obesity; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation Control Group (Active Comparator): Participants assigned to the psychoeducation control group will receive informational handouts about overweight and obesity, including current daily sleep, diet, and physical activity recommendations to prevent/treat overweight and obesity.
  Interventions: Other: Psychoeducation
- Emotion Regulation and Self-Monitoring Program (Experimental): Participants randomized to this condition will receive an active intervention which includes 4 weeks of an emotion regulation and self-monitoring program. Participants will attend telehealth group sessions once weekly and be asked to self-monitor their mood and health behaviors daily between sessions.
  Interventions: Behavioral: Emotion regulation and self-monitoring to treat pediatric obesity

INTERVENTIONS:
Behavioral: Emotion regulation and self-monitoring to treat pediatric obesity — Participants will attend telehealth group sessions once weekly and be asked to self-monitor their mood and health behaviors daily between sessions.
  Arms: Emotion Regulation and Self-Monitoring Program
Other: Psychoeducation — Participants who are randomized to the control group will receive an online, one-time, self-led psychoeducation program with information about current daily sleep, diet, and physical activity recommendations (e.g., information about sleep hygiene, the food pyramid, and recommendations for 60 minutes of moderate-to-vigorous physical activity daily).
  Arms: Psychoeducation Control Group

SUMMARY:
The goal of this clinical trial is to learn if an emotion regulation and self-monitoring intervention can help treat overweight and obesity in teens. The main question it aims to answer is:

* Does emotion regulation and self-monitoring help reduce biases in teens with overweight and obesity?
* Do changes in biases relate to changes in health functioning and health behavior?

Researchers will compare the intervention to the provision of educational handouts about overweight and obesity to see if the intervention is more effective.

Participants will:

* Complete self-report questionnaires, an fMRI scan, and have their blood drawn
* Received educational handouts or attend weekly telehealth group sessions weekly for four weeks and be asked to self-monitor their mood and behavior between sessions
* Return to complete the same questionnaires, fMRI and blood draw procedures

ELIGIBILITY:
Inclusion Criteria:

* Being English-proficient
* Ages 11-14
* At or above the 85th BMI percentile based on age and sex norms
* Having access to WIFI or cellular data to attend the telehealth groups
* Living in a home in Lubbock County (TX) or surrounding areas.

Exclusion Criteria:

* Having a psychiatric or medical diagnosis that interferes with participation (e.g., significant developmental delay; pregnancy)
* Current enrollment in overweight/obesity treatment.
* Because the study will include entering an MRI scanner, additional standard exclusion criteria will be considered (e.g., having immovable medical devices with batteries, body piercings on the head/face, and having substantial visual impairment that cannot be corrected with staff-provided glasses)

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage BOLD (Blood Oxygenation Level Dependent) signal change | From enrollment to the end of treatment at week 5
  Used to index pre-post changes in neuronal responsiveness to obesity-related cues
Glucose tolerance per blood samples | From enrollment to the end of treatment at week 5
  Used to index pre-post changes in health indicators linked to overweight and obesity severity
Triglycerides per blood samples | From enrollment to the end of treatment at week 5
  Used to index pre-post changes in health indicators linked to overweight and obesity severity
Cholesterol per blood samples | From enrollment to the end of treatment at week 5
  Used to index pre-post changes in health indicators linked to overweight and obesity severity
C peptide per blood samples | From enrollment to the end of treatment at week 5
  Used to index pre-post changes in health indicators linked to overweight and obesity severity
Emotion regulation per Difficulties in Emotion Regulation Scale-Short Form (DERS-SF) and Positive Affect (DERS-PA) versions | From enrollment to the end of treatment at week 5
  Used to index pre-post changes in difficulties with positive and negative emotion regulation. Sum scores and average scores for each measure and subscale are used, with higher scores indicating greater difficulties with each domain
Self-report disordered eating cognitions and behaviors per Eating Disorder Examination-Questionnaire | From enrollment to the end of treatment at week 5
  Used to index pre-post changes in health behavior. Items are summed together and averaged, with higher scores indicating greater disordered eating cognitions and behaviors
Self-report average daily minutes and intensity of physical activity per Patient-Reported Outcomes Measurement Information System (PROMIS) scale | From enrollment to the end of treatment at week 5
  Used to index pre-post changes in health behavior. Items are summed together with higher scores indicating greater frequency and intensity of physical activity
Self-report average daily minutes and intensity of physical activity per Physical Activity Questionnaire for Adolescents (PAQ-A) | From enrollment to the end of treatment at week 5
  Used to index pre-post changes in health behavior. Items are summed together with higher scores indicating greater frequency and intensity of physical activity
Self-report average daily minutes engaging in sedentary behavior per National Health and Nutrition Examination Survey (NHANES) items | From enrollment to the end of treatment at week 5
  Used to index pre-post changes in health behavior. Items are summed together with higher scores indicating more frequent sedentary behavior
Self-report acceptability per face-valid questionnaire | From enrollment to the end of treatment at week 5
  Sum scored, with higher score indication higher acceptability
Percentage of sessions attended (by participant) | From enrollment to study completion, an average of 1 year
  Used to index intervention feasibility
Number of participants enrolled | From enrollment to study completion, an average of 1 year
  Used to index intervention feasibility
Rate of attrition | From enrollment to study completion, an average of 1 year
  Used to index intervention feasibility

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be shared upon request and approval. To maintain privacy/confidentiality, fMRI scans and blood samples will not be shared, though specific values can be provided upon request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months.
Access Criteria: Access to IPD will can be requested by qualified researchers following review and approval of a research proposal, confirmation of IRB approval, and execution of a Data Sharing Agreement. For more information or to submit a request, please contact Dr. Caroline Cummings at carolicu@ttu.edu